CLINICAL TRIAL: NCT01085370
Title: Psychological Interventions in Children After Road Traffic Accidents or Burns: a Randomized Controlled Study
Brief Title: Psychological Interventions in Children After Road Traffic Accidents or Burns
Acronym: PICARTA-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PICARTA-B
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Acute Stress Disorder
Keywords: posttraumatic stress; prevention; children; acute stress disorder due to burn injury or injuries associated with road traffic accidents
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): standard medical care only
- Intervention group (Experimental): 2 sessions with early psychological interventions
  Interventions: Other: Early psychological intervention

INTERVENTIONS:
Other: Early psychological intervention — 3 modules: psychoeducation, reconstruction of the trauma, coping skills
  Arms: Intervention group

SUMMARY:
Within a randomized controlled design the effects of a brief early psychological intervention (child, parents) after road traffic accidents or burns shall be examined in a sample of 120 children and adolescents (aged 2 to 16 years). During the first seven days after the accident a screening for the risk of developing a posttraumatic stress disorder is conducted to divide the participants into a "high risk" and a "low risk" group. Participants with a low risk are excluded from the intervention study but reassessed six months after their accident to validate the screening instrument. After a baseline assessment within 14 days after the accident participants of the high risk group are randomly assigned to an intervention group (n = 60) or a control group (n = 60). The latter receive standard medical care. Children of the intervention group are provided with a brief age appropriate two-session intervention that includes a detailed reconstruction of the accident, psychoeducation and discussion of helpful coping strategies. Both the control and the intervention group are reassessed by blind raters at 3 and 6 months after the accident. Assessment of outcome includes measures of posttraumatic stress symptoms, depression, anxiety, behavior, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-16 years
* Glasgow Coma Scale (GCS) > 8
* German speaking
* Burn accident or road traffic accident

Exclusion Criteria:

* Glasgow Coma Scale (GCS) < 9
* more than 2 weeks in the Pediatric Intensive Care Unit
* no command of German
* previous mental retardation

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Clinician administered PTSD Scale for Children/Adolescents (CAPS-CA) and Child Posttraumatic Stress Disorder Semistructured Interview and Observational Scale (PTSDSSI) | Baseline, 3 months, 6 months post intervention

SECONDARY OUTCOMES:
KIDSCREEN-Questionnaire / TAPQOL-Questionnaire (health-related quality of life) | Baseline, 3 months, 6 months post intervention
Child behavior Child Behavior Checklist (CBCL) | Baseline, 3 months, 6 months post intervention
Child Depression Inventory (CDI) | Baseline, 3 months, 6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Markus A Landolt, PhD, Principal Investigator — University Children's Hospital Zurich, Psychosomatic and Psychiatry
Locations (1):
- Unviersity Children's Hospital, Psychosomatic and Psychiatry, Zurich, Switzerland

REFERENCES:
- [Derived] Kramer DN, Hertli MB, Landolt MA. Evaluation of an early risk screener for PTSD in preschool children after accidental injury. Pediatrics. 2013 Oct;132(4):e945-51. doi: 10.1542/peds.2013-0713. Epub 2013 Sep 23. PMID 24062371